CLINICAL TRIAL: NCT07206511
Title: Clinical Outcomes of Initially Unresectable Hepatocellular Carcinoma Patients Receiving TACE/HAIC Plus Anti-Angiogenic Agents and Immune Checkpoint Inhibitors as Conversion Therapy, Achieving Complete Radiological Response or Resectability, Followed by Systemic Treatment or Surgical Resection: A Prospective Cohort Study
Brief Title: Conversion Therapy Using TACE/HAIC With Anti-Angiogenic and Immunotherapy for Initially Unresectable Hepatocellular Carcinoma Achieving Complete Response or Resectability, Followed by Surgery or Continued Systemic Treatment: A Prospective Cohort Study
Acronym: THAI-CONVERT
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Jian Zhou, Hospital President, Shanghai Zhongshan Hospital
Other Study IDs: B2025-437R
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Unresectable Hepatocellular Carcinom
Keywords: Hepatocellular Carcinoma; Conversion Therapy; Radiological Complete Response; Systemic Therapy; Surgical Resection
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Systemic Therapy Group: Patients with initially unresectable hepatocellular carcinoma who achieved complete radiological response or resectability after TACE/HAIC + anti-angiogenic agents + immune checkpoint inhibitors and then continued systemic therapy.
- Surgical Resection Group: Patients with initially unresectable hepatocellular carcinoma who achieved complete radiological response or resectability after TACE/HAIC + anti-angiogenic agents + immune checkpoint inhibitors and then underwent surgical resection.

SUMMARY:
This is a prospective cohort study designed to evaluate the effectiveness and safety of two post-conversion treatment strategies for patients with initially unresectable hepatocellular carcinoma (uHCC). Participants first receive conversion therapy with transarterial chemoembolization (TACE) or hepatic arterial infusion chemotherapy (HAIC) combined with anti-angiogenic agents and immune checkpoint inhibitors (ICIs). After this therapy, patients who achieve complete radiological response (rCR) or meet resectability criteria will either undergo surgical resection or continue systemic therapy. The study aims to compare outcomes between these two strategies to help guide treatment decisions for advanced liver cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent.
2. Age 18-75 years.
3. Hepatocellular carcinoma (HCC) confirmed by histology/cytology or diagnosed according to the AASLD criteria.
4. Initially unresectable HCC (uHCC), defined according to the Chinese Guidelines for Diagnosis and Treatment of Primary Liver Cancer (2024 edition) and the Chinese Expert Consensus on Conversion and Perioperative Therapy for Primary Liver Cancer (2024 edition): HCC considered unsafe for curative resection due to inability to ensure both oncological completeness (R0 resection) and functional hepatic reserve (adequate future liver remnant with good vascular supply and biliary drainage to maintain postoperative liver function and minimize morbidity and mortality). Mainly includes CNLC stage Ib-IIIa or potentially resectable cases. Some stage Ia patients may also be considered uHCC if the tumor is adjacent to major intrahepatic vessels or involves the first/second hepatic hilum making R0 resection infeasible, or if severe cirrhosis increases risk of postoperative liver failure and complications; these can be considered after successful conversion and supportive treatment.
5. No prior systemic therapy before conversion treatment.
6. Conversion therapy regimen must include TACE or HAIC plus anti-angiogenic agents and immune checkpoint inhibitors (ICIs).
7. Anti-angiogenic agents may include lenvatinib, sorafenib, apatinib, donafenib, anlotinib, bevacizumab.
8. ICIs may include pembrolizumab, atezolizumab, nivolumab, sintilimab, tislelizumab, toripalimab, penpulimab, cadonilimab, KN-046.
9. After conversion therapy, hepatic lesions achieve radiological complete response (rCR) by mRECIST criteria on contrast-enhanced CT or MRI, or are assessed to have reached resectability criteria (eligible for curative hepatectomy or downstaging enabling safe surgery).
10. After achieving rCR or resectability, patients must have received either liver resection or continued systemic therapy with scheduled follow-up.
11. Child-Pugh class A or B liver function.
12. Eastern Cooperative Oncology Group performance status (ECOG PS) 0-1.

Exclusion Criteria:

1. Presence of another primary malignancy in other organs.
2. History of other malignancies.
3. Recurrent HCC occurring <2 years after previous curative surgery or adjuvant therapy.
4. Received treatments other than TACE or HAIC plus anti-angiogenic agents and ICIs during the conversion phase.
5. Received treatments during postoperative or maintenance systemic therapy that differ from the initial conversion regimen.
6. Severe organ dysfunction.
7. Incomplete radiological assessment data after treatment.
8. Child-Pugh class C liver function.
9. Pregnant or breastfeeding women.
10. Patients undergoing only functional future liver remnant (FLR) hypertrophy procedures (e.g., ALPPS or PVE) for insufficient FLR without other criteria for uHCC conversion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are adults (18-75 years) with initially unresectable hepatocellular carcinoma (uHCC) diagnosed by histology/cytology or according to AASLD criteria and Chinese national guidelines. These patients have received conversion therapy consisting of transarterial chemoembolization (TACE) or hepatic arterial infusion chemotherapy (HAIC) combined with anti-angiogenic agents and immune checkpoint inhibitors (ICIs). After conversion therapy, participants have achieved radiological complete response (rCR) or reached resectability criteria and then either undergo curative liver resection or continue systemic therapy. Eligible patients must have Child-Pugh class A or B liver function and ECOG performance status 0-1.
Sampling Method: Non-Probability Sample
Enrollment: 278 (Estimated)
Dates: Start 2025-10-09 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Event-Free Survival (EFS) | From initiation of post-conversion therapy to the first documented event (recurrence, progression, or death), up to 36 months
  Defined as the time from the date of achieving rCR or resectability criteria to the time of becoming inoperable, recurrence, progression, or death from any cause for uHCC patients.

SECONDARY OUTCOMES:
2-Year Event-Free Survival (EFS) Rate | 2 years after initiation of post-conversion therapy
  Defined as the rate of no events (recurrence, progression, or death from any cause) occurring in rCR patients over 2 years.
Overall Survival (OS) | Up to 36 months after initiation of post-conversion therapy
  Defined as the survival time from the day of achieving rCR to death from any cause。
Treatment Safety | From initiation of post-conversion therapy through 30 days after last treatment or surgery, up to 36 months follow-up
  : The incidence of adverse events in the surgery group and the systemic therapy group. Adverse events recorded on the CRF will be mapped to preferred terms using the Medical Dictionary for Regulatory Activities (MedDRA). Severity, seriousness/grade, and the relationship with the study treatment will be assessed by the investigators. The seriousness/grade will be defined according to the National Cancer Institute (NCI) CTCAE v5.0.
Cost-Effectiveness of Post-Conversion Treatment Strategies | Up to 36 months after initiation of post-conversion therapy
  The cost-effectiveness ratio (C/E) is defined as the ratio of time to an event (EFS) or overall survival (death) from rCR to all direct costs (medical expenses, including outpatient and inpatient), and will be compared between the two groups.

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-08): https://cdn.clinicaltrials.gov/large-docs/11/NCT07206511/Prot_SAP_000.pdf